CLINICAL TRIAL: NCT01875146
Title: Effects of High-intensity Interval Training in Combination With Side-alternating Whole-body Vibration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: vyc
Record Dates: First submitted 2013-05-16; First posted 2013-06-11 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-12

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

ARMS (4):
- 4x4 min HIT (Active Comparator): Conventional 4x4 min high-intensity interval training
  Interventions: Other: 4x4 min HIT
- 4x4 min HIT + WBV (18 Hz) (Experimental): 4x4 min high-intensity interval training in combination with whole-body vibration at 18 Hz during the active rest
  Interventions: Other: 4x4 min HIT + WBV (18 Hz)
- 4x4 min HIT + WBV (30 Hz) (Experimental): 4x4 min high-intensity interval training in combination with whole-body vibration at 30 Hz during the active rest
  Interventions: Other: 4x4 min HIT + (30 Hz)
- whole-body vibration at 30 Hz (Active Comparator): 4x3 min whole-body vibration at 30 Hz
  Interventions: Other: whole-body vibration at 30 Hz

INTERVENTIONS:
Other: 4x4 min HIT — Conventional 4x4 min high-intensity interval training
  Arms: 4x4 min HIT
Other: 4x4 min HIT + WBV (18 Hz) — 4x4 min high-intensity interval training in combination with whole-body vibration at 18 Hz during the active rest
  Arms: 4x4 min HIT + WBV (18 Hz)
Other: 4x4 min HIT + (30 Hz) — 4x4 min high-intensity interval training in combination with whole-body vibration at 30 Hz during the active rest
  Arms: 4x4 min HIT + WBV (30 Hz)
Other: whole-body vibration at 30 Hz — 4x3 min whole-body vibration at 30 Hz
  Arms: whole-body vibration at 30 Hz

SUMMARY:
Investigation of the training effects following 8 weeks of high-intensity interval training (HIT)in combination with side-alternating whole-body vibration compared to conventional HIT or side-alternating whole-body vibration. The adaptations are investigated on a molecular (muscle biopsy of the M. vastus lateralis) and systemic (e.g. cycling, jumping mechanography, dynamometry) level. In addition, the acute effects of the first and last training session will be investigated on a molecular (e.g. satellite cell activation, mRNA abundance) and systemic (e.g. ventilatory ga exchange, heart rate, rating of perceived exertion) level.

ELIGIBILITY:
Inclusion criteria: - male

* no fever / no common cold at the beginning of the study
* between 18 and 35 years of age
* non-smoker
* no known cardiovascular or orthopedic problems
* no cardiac pacemaker
* fullfills healts questionnaire's requirements

Exclusion criteria: - female

* fever / common cold at beginning of study
* age under 18 oder above 35y
* smoker
* cardiovascular or orthopedic problems
* cardiac pacemaker
* does not fullfill health questionnaire's requirements

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Critical Power | 8 weeks intervention
  The differences in changes in Critical Power [Watts] are compared between the 4 training groups. For this purpose, participants complete before and after the training intervention an incremental cycling ramp test and 4 cycling constant-load tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hans H Jung, Prof MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Mueller SM, Aguayo D, Zuercher M, Fleischmann O, Boutellier U, Auer M, Jung HH, Toigo M. High-intensity interval training with vibration as rest intervals attenuates fiber atrophy and prevents decreases in anaerobic performance. PLoS One. 2015 Feb 13;10(2):e0116764. doi: 10.1371/journal.pone.0116764. eCollection 2015. PMID 25679998